CLINICAL TRIAL: NCT03991247
Title: Evaluation of Psychosomatic Spa Treatment With Crenotherapy to Potentiate the Implementation of Behavioral Measures for Insomnia Disorder Management
Brief Title: Evaluation of Spa Treatment on Insomnia
Acronym: SOMNOTHERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: University Hospital, Bordeaux (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2018-01; 2019-A00043-54 (Other: ANSM Number (ID-RCB))
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Insomnia
Keywords: Spa treatment; Cognitive Behavioral Therapy; Internet delivered self-help program; Insomnia; Sleep restriction; stimulus control; crenotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Behavioral therapy program + spa therapy (Experimental): Patient following a program of computerized behavioral therapy for insomnia management during a 3 weeks spa treatment.
  Interventions: Behavioral: Computerized behavioral therapy program delivered by internet for insomnia management; Other: Spa treatment
- Internet Behavioral therapy program at home (Active Comparator): Patient following a program of computerized behavioral therapy for insomnia management during 3 weeks at home.
  Interventions: Behavioral: Computerized behavioral therapy program delivered by internet for insomnia management

INTERVENTIONS:
Behavioral: Computerized behavioral therapy program delivered by internet for insomnia management — The online program consists in restriction of time in bed and stimulus control instructions.
  First, patient will complete an on-line sleep diary during 2 weeks. The personalized program is then activated by a practitioner (phone interview) who both assesses restriction of time in bed and delivers instructions of stimulus control. Then, restriction of time in bed is administered by the internet-delivered self-help program. The participant still completes his on-line sleep diary every day. Every 7 days, according mean sleep efficiency, a new sleep schedule recommendation is given to the participant. In addition, the program delivers everyday a set of instructions (stimulus control) designed to re-associate the bed/bedroom with sleep and to re-establish a consistent sleep wake schedule. The duration of restriction of time in bed program is 3 weeks (during spa treatment or at home depending on the allocated arm).
Other: Spa treatment — Spa treatment is harmonized in the different stations. It consists in:
  * a medical thermal follow-up: weekly medical consultation of 15 minutes during the 3 weeks spa treatment.
  * an institutional follow-up: support, help and monitoring of patients during spa treatment
  * Crenotherapy: 18 baths of 10 minutes in running water, 18 spa showers of 3 minutes, 9 massages under water of 20 minutes, 18 baths of 10 minutes in pool. Water temperature of pool is between 31°C and 33°C. Water temperature for other care is 35°C and 38°C.
  Arms: Internet Behavioral therapy program + spa therapy

SUMMARY:
Persistant insomnia is a common sleep disorder that affects approximately 20% of the French population. The standard treatment for chronic insomnia is Cognitive-Behavioral Therapy (CBT).

Behavioral measures can be difficult to implement for the patient alone at home.

Spa therapy with psychosomatic orientation allows to implement hygiene rules and structure rhythms of life. In addition, recent studies have shown that spa treatment, including crenotherapy, is effective in somatic complaints related to anxiety and benzodiazepine withdrawal.

The spa treatment could therefore provide ideal conditions for the implementation of behavioral measures for insomnia management.

The objective of SOMNOTHERM study is to measure efficiency on insomnia complaints at 8 weeks of a the implementation of a Behavioral therapy program for insomnia delivered by an internet software combined to a spa treatment compared to implementation of the same program at home (standard care).

DETAILED DESCRIPTION:
Persistant insomnia is a common sleep disorder that affects approximately 20% of the French population.

The standard treatment for chronic insomnia is Cognitive-Behavioral Therapy (CBT). This therapy is based on 4 components: sleep restriction, stimulus control, cognitive therapy and sleep hygiene education. Unfortunately, there are an insufficient number of trained CBT experts especially in France.

Online programs based on CBT principles (e-CBT) have been proved to be effective in improving the sleep and daytime functioning in this population. Thus e-CBT can be an effective alternative to conventional CBT.

Behavioral measures, however, remains difficult for patients to implement alone at home.

Spa therapy with psychosomatic orientation allows to implement hygiene rules and structure rhythms of life. In addition, recent studies have shown that spa treatment, including crenotherapy, is effective in somatic complaints related to anxiety and benzodiazepine withdrawal.

In this context, spa treatment with psychosomatic orientation appears conducive to implement hygiene rules and structure rhythms of life. The spa treatment could therefore provide ideal conditions for the implementation of behavioral measures of insomnia management (sleep hygiene, stimulus control and time in bed restriction) and could have a very beneficial effect on persistent insomnia disorder.

This non-pharmacological therapy could also reduce hypnotics consumption (especially benzodiazepine).

The main hypothesis of the study is that behavioral measures of insomnia management delivered by an internet software program combined to a spa treatment will be more effective on insomnia complaints (evaluated at 8 weeks) than the same program implemented at home.

Patients will be followed during 6 months after the beginning of the program. Subjects' recruitment will be carried out from the list of patients registered for a spa treatment in one of the five spa centers participating in the study (Les Thermes de Saujon, Les Grands Thermes de Bagnères de Bigorre, Les Thermes de Divonne-les-Bains, Les thermes de Néris-les-Bains, Les Thermes d'Ussat-les-Bains).

Study visits will be conducted by the coordinating center (CHU Bordeaux) by telephone interviews or video calls with participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 80 years old
* Registered at one of the participating spas, for a psychosomatic spa treatment scheduled for the next 12 months, but within a period of more than 16 weeks.
* ISI score ≥ 8 on the pre-selection questionnaire
* Person with a persistent insomnia disorder, with or without comorbidities, according to DSM 5
* Owning or having access to a computer / tablet or smartphone and to an internet connection
* Affiliated to a national health service
* Having given written informed consent to participate in the trial.

Exclusion Criteria:

* Strong suspicion of obstructive sleep apnea (OSA) syndrome on the STOP-BANG questionnaire and restless legs syndrome on the RLS screening questionnaire
* Having started antidepressant treatment in the last 2 months or whose treatment dose has been increased in the last 2 months
* Having started treatment with anxiolytic, hypnotic or neuroleptic in the last month or whose dosage of treatment has been increased in the last month
* Having carried out a spa treatment in the last 6 months, whatever the specialty.
* Registered to follow a complementary program for insomnia disorders during the planned spa treatment
* Pregnant or lactating women
* Major under guardianship or curatorship
* Night and shift-workers
* Having undertaken trans-meridian travel (± 3H) in the previous 1 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Scale (ISI) score | Week 10 = 8 weeks after beginning of computerized behavioral therapy (starting of time in bed restriction)
  7-item questionnaire assessing insomnia nature, severity and impact. The global score ranges from 0 to 28.

SECONDARY OUTCOMES:
Total sleep time (TST) obtained by sleep diary | Every night between starting of sleep diary completion (Day 0) and Month 6 (study termination)
  Total sleep time = total sleep episode minus awake time. Subject records in his online sleep diary bedtime, wake-up time, time asleep, intra-night awakenings.
Sleep efficiency (SE) obtained by sleep diary | Every night between starting of sleep diary completion (Day 0) and Month 6 (study termination)
  Ratio of total sleep time (TST) to time in bed (TIB) (multiplied by 100 to yield a percentage).
  Subject records in his online sleep diary bedtime, wake-up time, time asleep, intra-night awakenings.
Sleep latency obtained by sleep diary | Every night between starting of sleep diary completion (Day 0) and Month 6 (study termination)
  Length of time to accomplish the transition from full wakefulness to sleep. Subject records in his online sleep diary bedtime, wake-up time, time asleep, intra-night awakenings.
Insomnia Severity Scale (ISI) score | On Day 0, Week 5, Week 7, Month 4, Month 6
  7-item questionnaire that assesses insomnia nature, severity and impact.
EQ-5-D | On Day 0, Week 5, Week 7, Week 10, Month 4, Month 6
  Standardized instrument for measuring generic health status.
The Presleep State Arousal Scale (PSAS) | On Day 0, Week 5, Week 7, Week 10, Month 4, Month 6
  16-item questionnaire assessing whether the respondent experienced somatic (8 items, eg heart rate) or cognitive hyperarousal (eg racing thoughts) at bedtime
Hospital Anxiety and Depression Scale (HAD) | On Day 0, Week 5, Week 7, Week 10, Month 4, Month 6
  14-item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.
Short Version of the Functional Outcomes of Sleep Questionnaire (FOSQ) | On Day 0, Week 5, Week 7, Week 10, Month 4, Month 6
  10 item questionnaire assessing the impact of excessive sleepiness on activities of daily living
Rate of discontinuation and rate of reduction of anxiolytic hypnotic drugs and hypnotics | On Day 0, Week 5, Week 7, Week 10, Month 4, Month 6
  Every day anxiolytic hypnotic drugs and hypnotics daily dose
Acceptability E-scale (AES) | On week 10 (after computerized behavioral therapy program)
  6-item self-reported questionnaire that evaluates the extent to which patients find E-health systems acceptable
Client Satisfaction Questionnaire (CSQ-8) | On week 10 (after computerized behavioral therapy program)
  8-item questionnaire easily scored and administered measurement that is designed to measure client satisfaction with services.
Sleep Condition Indicator (SCI) | On Day 0
  brief 8-item scale which measures sleep problems against the DSM-5 criteria for insomnia disorder
The Pittsburgh Sleep Quality Index (PSQI) | On Day 0
  self-report questionnaire that assesses sleep quality over a 1-month time interval
Cognitive Scale of Attachment to Benzodiazepines ("Echelle cognitive d'attachement aux benzodiazépines" ECAB) | On Day 0
  10-item scale assessing cognitive component of attachment to benzodiazepines
The Munich ChronoType Questionnaire (MCTQ) | On Day 0
  Questionnaire to determine Chrono Type.
The Epworth Sleepiness Scale (ESS) | On Day 0
  8-item questionnaire assessing daytime sleepiness
Freiburg Mindfulness Inventory - short version (FMI) | On Day 0
  questionnaire for measuring mindfulness
Krueger's personality inventory for DSM-5 in its brief form (PID-5-BF) | On Day 0
  25-item self-report questionnaire assessing the presence and severity of the five maladaptive personality traits outlined in DSM-5.
The Arousal Predisposition Scale (APS) | On Day 0
  12-item questionnaire assessing whether the respondent considers her/himself a stressful and emotionally reactive person
The Ford Insomnia to Stress Scale (FIRST) | On Day 0
  9-item questionnaire assessing whether past and future stressful events are likely to affect sleep quality
The "locus of control for technology"-questionnaire ("Kontrollüberzeugungen im Umgang mit Technik" - KUT) | On Day 0
  8-item questionnaire assessing the specific interaction with technical environments of users

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
Patient could request investigator or Data Protection Officer an access to IPD according to French regulation (act No. 78-17 of 6 January 1978 on data processing, data files and individual liberties, amended by act No. 2004-801 of 6 August 2004) and he EU General Data Protection Regulation (GDPR) of 27 april 2016 applicable since 25 May 2018.